CLINICAL TRIAL: NCT01547533
Title: Study of Benznidazole Transfer Into Breastmilk in Lactating Women Treated for Chagas Disease
Brief Title: Study of Benznidazole Transfer Into Breastmilk in Lactating Women With Chagas Disease
Acronym: LACTBENZ
Status: Completed | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Facundo Garcia-Bournissen, Associate Researcher, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: LACT-BENZNIDAZOLE
Record Dates: First submitted 2012-03-01; First posted 2012-03-08 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Chagas Disease; Lactation
Keywords: Chagas disease; lactation; breastmilk; postpartum period; infants; pediatric clinical pharmacology; developmental clinical pharmacology; parasitology; trypanosoma cruzi
MeSH Terms: conditions — Chagas Disease; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breastmilk; plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lactating Women with Chagas disease: Women with Chagas disease who fulfill clinical criteria for treatment with benznidazole, and who are also lactating

SUMMARY:
The investigators propose to study the transfer of benznidazole into breastmilk from the blood of lactating women who receive the drug for the treatment of Chagas disease. Breastmilk and blood samples will be obtained from these patients at given times after they take the clinically indicated medication, and the concentrations in both matrices will be compared to estimate degree of transfer, which in turn will be used to evaluate potential degree of exposure of infants breastfed by these women. This study will help clarify safety of continuing breastfeeding while receiving treatment with benznidazole for Chagas disease.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women with Chagas disease, not treated before
* Use of contraception

Exclusion Criteria:

* History of allergy to benznidazole or its excipients
* Pregnancy
* Significant heart involvement (due to Chagas disease)
* Significant systemic diseases that could affect the interpretation of the results in the opinion of the principal investigator

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: population of young women with Chagas disease referred to our center for evaluation and treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Benznidazole concentration in breastmilk and in plasma | at randomly selected time points during the 30 days of treatment
  Randomly obtained breastmilk samples will be obtained to both evaluate the breastmilk / plasma concentration ratio of the drug, and to develop a population pharmacokinetics model of drug trasfer into breastmilk, if possible.
  Breastmilk concentrations will be used to calculate potential infant exposure through breastmilk to the medication (benznidazole) taken by the mother

SECONDARY OUTCOMES:
incidence of adverse drug reactions in women treated with benznidazole during lactation | throughout the 30 days of treatment
  Women receiving treatment with benznidazole while lactating, enrolled in the study will be followed according to current clinical guidelines, and monitored during the 60 days of the treatment (as per Chagas disease treatment guidelines), and monthly for 3 months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Facundo Garcia Bournissen, MD PhD, Principal Investigator — Buenos Aires Children´s Hospital Ricardo Gutierrez ; CONICET
Locations (1):
- Parasitology and Chagas Service, Buenos Aires Children´s Hospital Ricardo Gutierrez, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Garcia-Bournissen F, Moroni S, Marson ME, Moscatelli G, Mastrantonio G, Bisio M, Cornou L, Ballering G, Altcheh J. Limited infant exposure to benznidazole through breast milk during maternal treatment for Chagas disease. Arch Dis Child. 2015 Jan;100(1):90-4. doi: 10.1136/archdischild-2014-306358. Epub 2014 Sep 10. PMID 25210104